CLINICAL TRIAL: NCT05441111
Title: Combining Guided Self-help Approaches for Common Mental Disorders
Brief Title: Low-intensity Stepped Care for Internalizing Distress
Acronym: COMET-DWM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Lorenzo Lorenzo-Luaces, Assitant Professor Pyschological and Brain Sciences, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11997
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Depression; Anxiety; Emotion Regulation
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMET + guided self-help bibliotherapy (Experimental): Participants are given access to a single session intervention the Common Elements Toolbox (COMET) and, a week after, are given access to the World Health Organization's (WHO) "Doing what matters in times of stress: An illustrated guide" (https://www.who.int/publications/i/item/9789240003927) virtually (i.e., as a pdf) and/or in print. Each participant is assigned an "eCoach" -- an undergraduate, post-baccalaureate, or graduate research assistant -- who will meet with the participant for a 60-minute welcome call describing the intervention and 3-6 sessions of guidance focused on promoting adherence to the manual and using skills in everyday life.
  Interventions: Behavioral: Common Elements Toolbox; Behavioral: Doing What Matters in Times of Stress: An Illustrated Guide; Behavioral: Guided self-help
- COMET + unguided self-help bibliotherapy (Active Comparator): Participants are given access to a single session intervention the Common Elements Toolbox (COMET) and, a week after, are given access to the World Health Organization's (WHO) "Doing what matters in times of stress: An illustrated guide" (https://www.who.int/publications/i/item/9789240003927) virtually (i.e., as a pdf) and/or in print. Participants are left to read the book on their own (i.e., without an eCoach)
  Interventions: Behavioral: Common Elements Toolbox; Behavioral: Doing What Matters in Times of Stress: An Illustrated Guide

INTERVENTIONS:
Behavioral: Common Elements Toolbox — COMET consists of the following modules: cognitive restructuring (labeled "flexible thinking"), behavioral activation (labeled "positive activities"), gratitude, and self-compassion. Participants complete these COMET modules by themselves. The format is reading psychoeducational along with completing specific activities
  Other Names: COMET; Single-session intervention
Behavioral: Doing What Matters in Times of Stress: An Illustrated Guide — From the WHO's website: Doing What Matters in Times of Stress: An Illustrated Guide is a stress management guide for coping with adversity. The guide aims to equip people with practical skills to help cope with stress. A few minutes each day are enough to practice the self-help techniques. The guide can be used alone or with the accompanying audio exercises.
  Informed by evidence and extensive field testing, the guide is for anyone who experiences stress, wherever they live and whatever their circumstances.
  Other Names: Self-help Plus
Behavioral: Guided self-help — Participants in the guided self-help condition are assigned an "eCoach" who provides emotional support as well as who promote adherence to the intervention
  Arms: COMET + guided self-help bibliotherapy

SUMMARY:
The purpose of this study is to test the feasibility and efficacy of combining a single session intervention, COMET, with a self-help intervention, Doing what matters in times of stress. In step I, all individuals receive COMET. In Step II, all individuals receive Doing what matters in times of stress but are randomized 1:1 to guided (Doing what matters in times of stress with paraprofessional support) vs. unguided self-help (Doing what matters in times of stress with no support).

DETAILED DESCRIPTION:
The first page participants will see is the informed consent document describing the study, delineating risks/benefits, payment, who to contact with problems, etc. Once participants have read through the informed consent, those who wish to participate will be taken to the survey battery.

The baseline survey should take about 15 minutes to complete. Individuals who score at least a 6 on the Kessler Psychological Distress Scale (K6) are eligible to participate. After participants are deemed eligible, they will be randomized to one of 2 conditions: guided self-help bibliotherapy or unguided self-help bibliotherapy. Participants who qualify and are randomized to the guided self-help condition will provide their phone number, email, address, whether they would like the Doing what matters in times of stress book to also be mailed to them, what their preferred method of initial contact is, and a list of timeframes in which they would have the privacy to be contacted by the research team. Participants who qualify and are randomized to the unguided self-help condition will provide their phone number, email, address, and confirm whether they would like the Doing what matters in times of stress book to also be mailed to them. Participants who do not qualify will be thanked for their time and receive the link to the book so they can use it on their own time if they wish.

After filling out their contact information, eligible participants will be taken directly to the Common Elements Toolbox (COMET) intervention. The COMET intervention will be delivered via Qualtrics and will include the following modules: cognitive restructuring (labeled "flexible thinking"), behavioral activation (labeled "positive activities"), gratitude, and self-compassion. The total time for completing the COMET intervention is around 45 minutes, which means the total approximate time for completing the entire baseline assessment (survey + COMET) is around 60 minutes.

For participants in the guided self-help condition, within 1 week of completing the baseline assessment a member of the research team will either email participants to schedule a time to call, or call eligible participants to explain the study in more detail, and answer any questions they may have. Participants will be sent a welcome email with the Doing what matters in times of stress book, a copy of the informed consent, and a participation guide. Each participant will receive a unique Zoom Health link to use for participation. These calls will not be recorded. This initial call will also serve to introduce the participant to the Doing what matters in times of stress book, create a plan for using the book, and schedule the remaining calls. The welcome call should take up to 30 minutes.

For participants in the unguided condition, within 1 week of completing the baseline assessment they will be emailed a copy of the book, the informed consent statement, the Making a Plan Worksheet, and a participation guide.

The next phase of the study involves participants using the Doing what matters in times of stress book either on its own or with guided interaction over video or phone calls. Each participant in the guided condition will meet weekly with a Research Assistant (RA) who will be trained to the therapeutic material and supportive accountability model. The supportive accountability model frames the relationship in self-help treatments as one in which the helper facilitates the participant's acquisition of skills by being supportive and promoting adherence to the material. This is different than the working alliance in individual therapy in which the patient and therapist work together on a mutually agreed-upon goal in that the relationship in guided self-help puts the emphasis on participants working on their own goals. To be clear, the RA will not be acting as a therapist - their role is only to help participants read through the book. The goal of these weekly guided interactions will be to provide supportive accountability and promote adherence to the intervention. The guided interactions will focus on how the participant interacts with the self-help material (i.e. how the participant feels about the material, goal setting, and performance monitoring). Guidance in the context of self-help has proven to increase treatment adherence compared to unguided self-administered treatment. This weekly guided self-help will be provided for 6 weeks. During this time the participant and trained RA will meet once a week for 3-6 weeks (depending on what the participant prefers). We will send out a reminder email the day before each meeting. Participants in the unguided condition will follow the same procedures, except they will not receive guidance.

ELIGIBILITY:
Inclusion Criteria:

* At least mild distress: K6 score ≥ 6
* Having reasonably regular access to the internet or a telephone

Exclusion Criteria:

* Suicidality: on the Patient Health Questionnaire 9 (PHQ9) item 9 ("thoughts that you would be better off dead, or of hurting yourself ") ≥ 2 ("more than half the days")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
6-week change in Kessler 6 Psychological Distress Scale (K6) | 6 weeks
  Changes in K6 from baseline to Week 6. The K6 is a measure of distress and the measure is scored on a scale of 0 - 24 where higher scores indicate higher distress (i.e., are negative). Thus, lower scores relative to baseline indicate more positive outcomes.
6-week change in the WHO 5 Well-being Index (WHO-5) | 6 weeks
  Changes in WHO-5 from baseline to Week 6. The WHO-5 is a measure of well-being and the measure is scored on a scale of 0 - 100 where higher scores indicate higher satisfaction with life (i.e., are positive). Thus, higher scores relative to baseline indicate more positive outcomes.

SECONDARY OUTCOMES:
6-week change in Emotion Regulation Scale (ERQ) - Reappraisal subscale | 6 weeks
  Changes in the ERQ Reappraisal subscale from baseline to Week 6. The Reappraisal scale is a measure of regulating emotions by engaging in reappraisal (i.e., changing the one one thinks about an emotion evoking stimuli), widely considered an adaptive strategy. The measured is scored on a 1-7 scale where higher scores indicate greater use of adaptive emotion regulation strategies (i.e., positive). Thus, higher scores relative to baseline indicate more positive outcomes.
6-week change in the Emotion Regulation Scale (ERQ) - Suppression subscale | 6 weeks
  Changes in the ERQ Suppression Scale from baseline to Week 6. The ERQ Suppression scale is a measure of regulating emotions by engaging in suppression (i.e., trying not to think or feel), which is considered a maladaptive emotion regulation strategy. The measure is scored on a scale of 1 - 7 where higher scores indicate higher use of suppression (i.e., negative). Thus, lower scores relative to baseline indicate more positive outcomes.
3-month change in Kessler 6 Psychological Distress Scale (K6; 0 - 24) | 3 months
  Changes in K6 from baseline to 3 months after the termination of the study. The K6 is a measure of distress and the measure is scored on a scale of 0 - 24 where higher scores indicate higher distress (i.e., negative). Thus, lower scores relative to baseline indicate more positive outcomes.
3-month change in the WHO 5 Well-being Index (WHO-5) | 3 months
  Changes in WHO-5 from baseline to 3 months after the termination of the study. The WHO-5 is a measure of well-being and the measure is scored on a scale of 0 - 100 where higher scores indicate higher satisfaction with life (i.e., are positive). Thus, higher scores relative to baseline indicate more positive outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon request.